CLINICAL TRIAL: NCT04094987
Title: Investigation of the Effect of Interfacial Pressure on Block Success During Anterior Quadratus Lumborum Block Application
Brief Title: Interfascial Pressure Into Ultrasound Guided Anterior Quadratus Lumborum Block Application
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bursa Yuksek Ihtisas Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Korgün Ökmen, Principal Investigator, Bursa Yuksek Ihtisas Training and Research Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2011-KAEK-25 2019/05-26
Record Dates: First submitted 2019-09-11; First posted 2019-09-19 (Actual); Last update posted 2021-02-02 (Actual); Status verified 2021-02

CONDITIONS: Block
MeSH Terms: conditions — Bites and Stings

STUDY DESIGN:
Intervention Model Description: prospective, cohort
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Quadratus Lumborum block (Experimental): We will use the ultrasound guided anterior Quadratus Lumborum Block.A peripheral nerve block catheter will be placed between the quadratus lumborum muscle and the psoas muscle with ultrasound
  Interventions: Device: inter-fascial pressure

INTERVENTIONS:
Device: inter-fascial pressure — The pressure between the fascia and the pressure line added to the catheter tip will be measured.

SUMMARY:
The block has been shown to be the result of abdominal analgesia as a result of application between the quadratus lumborum (QL) muscle and the leaves in the thoracolumbar fascia.

In this block, local anesthetic drugs are administered between the quadratus lumborum (QL) muscle and the anterior leaf in the thoracolumbar fascia.

In this way, it has been reported that it provides a good analgesia as it relieves somatic pain better in upper and lower abdominal surgeries.

DETAILED DESCRIPTION:
The mechanism of QLB analgesic contains many theories. This study includes the research relationship between the effect of fascial pressure and the success of the association block. We will use the ultrasound guided anterior Quadratus Lumborum Block. A peripheral nerve block catheter will be placed between the quadratus lumborum muscle and the psoas muscle with ultrasound.The pressure between the fascia and the pressure line added to the catheter tip will be measured.A peripheral nerve block catheter will be placed between the quadratus lumborum muscle and the psoas muscle with ultrasound. The pressure between the fascia and the pressure line added to the catheter tip will be measured.

ELIGIBILITY:
Inclusion Criteria:

Patients who were in the American Society of Anesthesiologists (ASA) I-III class

• Underwent laparoscopic cholecystectomy

Exclusion Criteria:

* Previous history of preoperative opioid use,
* Allergy to local anesthetics,
* The presence of any systemic infection,
* Uncontrolled arterial hypertension,
* Uncontrolled diabetes mellitus
* Presence of infection in the block area,

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2019-09-29 (Actual); Primary Completion 2019-10-15 (Actual); Study Completion 2020-09-15 (Actual)

PRIMARY OUTCOMES:
Interfascial Pressure (mm/hg) | 24 hours.
  İnterfascial pressure will be measured the postoperative 24. hours through catheter.

SECONDARY OUTCOMES:
sensory block level | peroperative 3 hours
  After the application, the sensory block level at the 30 minutes after the block application and 30 minutes after the operation will be determined by cold test.
Visual Analog Scale | Postoperative 24 hours
  Visual Analog Scale was used for pain.Pain intensity was measured using 0-10 cm visual analogue scale (VAS). (0=no pain, 10=intolerable pain)
analgesic use | Postoperative 24 hours
  analgesic use

CONTACTS AND LOCATIONS:
Overall Officials: Korgün Ökmen, Principal Investigator — Bursa Yuksek Ihtisas Training and Research Hospital
Locations (1):
- University of Health Sciences, Bursa Yuksek Ihtisas Training and Research Hospital, Bursa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No